CLINICAL TRIAL: NCT05906927
Title: Telemedicine for Home-based Management of Patients With Chronic Kidney Diseases and Comorbidities: Analysis of Current Models and Design of Innovative Strategies to Improve Quality of Care and Optimise Resource Utilization
Brief Title: Telemedicine for Home-based Management of Patients With Chronic Kidney Diseases and Comorbidities (NET-2018-12367206)
Acronym: Telemechron
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Azienda USL Toscana Nord Ovest (Other)
Responsible Party: Principal Investigator, Roberto Bigazzi, Emeritus Director of Operational Unit of Nephrology and Dialysis, Azienda USL Toscana Nord Ovest
Other Study IDs: Telemechron WP1-40/2019
Record Dates: First submitted 2023-03-02; First posted 2023-06-18 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is aimed to analyze the current models and to design innovative strategies to improve quality of care and optimise resource utilization of telemedicine (TM) in home-based management for the global care of patients with chronic kidney diseases (CKD). The main focus is on the prevention of complications, recurrence of unstabilization and optimal therapy for the global management of chronic pts through TM and e-Health. Reducing avoidable/unnecessary hospitalisation of pts with chronic conditions, through the effective implementation of a health care network, offering integrated care programs and applying chronic disease management models, should ultimately contribute to the improved efficiency of health systems.

DETAILED DESCRIPTION:
The investigators will design, test and evaluate innovative models for applying TM to the management of pts with chronic kidney diseases .

New models will be characterized by the followings:

* flexible adaptation to pts subgroups/ individual pts characteristics, including pts (and caregivers) expectation and willingness to participate actively in the process of care
* identification of technical components which are essential, accessory, useful or futile for different pts subgroups, including evaluation of pts abilities and preferences.
* definition of the team of care and the roles and responsibilities of each components: case manager, clinical manager etc
* pre-definition of outcome measures, that should include at least the evaluation of quality of life, perceived quality of care by the pts and caregivers, number and duration of hospitalizations.
* definition of Quality Assurance (QA) derived indicators related to risk and performance of TM implementation where needed

Finally, the investigators will collect a set of data allowing to analyse and validate the care model and to measure the patient adherence to the care plan as well as measure the performance of the predictive models based on this data.

ELIGIBILITY:
Inclusion Criteria for Peritoneal dialysis (PD) patients:

* patients already on treatment both in continuous home peritoneal dialysis (CAPD) and patients in nocturnal automated peritoneal dialysis (IPD)
* autonomous in their management of dialysis therapy,
* absence of acute or rapidly disabling comorbidities,
* ability to use a smart phone,
* home covered by fast optical fiber

Inclusion Criteria for Hemodialysis (HD) patients:

* Patients already in treatment, autonomous in their management of home dialysis therapy, or in dialysis at peripheral centers where the continuous presence of the nephrologist is not guaranteed
* Absence of acute or rapidly disabling comorbidities,
* Presence of a stable and well-functioning vascular access for hemodialysis,
* Ability to use a smart phone,
* Home covered by fast optical fiber

Inclusion Criteria for Chronic nephropathic patients undergoing predialysis:

* Patients already taken care of by the facility,
* Absence of acute or rapidly disabling comorbidities,
* Ability to use a smart phone,
* Home covered by fast optical fiber

Exclusion Criteria:

* History of malignant hypertension or accelerated hypertension within 6 months prior to study entry.
* History of drugs i.v. or alcohol abuse. History of cocaine abuse will be an exclusion criterion.
* Serious systemic disease that could affect the survival or course of the kidney disease.
* Body mass index greater than 35 Kg/m2 in men and 33 Kg/m2 in women. BMI is calculated as weight (kg)/height (m2).
* Myocardial infarction or cerebrovascular accident in the past 6 months
* Pregnancy or likelihood of becoming pregnant during the study period.
* Using nonsteroidal anti-inflammatory drugs (NSAIDs) for more than 1 week/month, excluding baby aspirin.
* Suspect that the participant will not be able to meet the protocol visits schedule.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We propose to consider 3 case studies: 2 patients on peritoneal dialysis , 2 patients on home hemodialysis and 4 patients attending pre-dialysis clinic .
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline number of days of hospitalization at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline number of days of hospitalization and the ones at 6 and 12 months will be performed. Data will be extracted from the data flows of healthcare information systems
Change from baseline number of home visits by the doctor at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline number of home visits by the doctor and the ones at 6 and 12 months will be performed. Data will be extracted from the data flows of healthcare information systems
Change from baseline number of doctor's office visits at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline number of doctor's office visits and the ones at 6 and 12 months will be performed. Data will be extracted from the data flows of healthcare information systems
Change from Baseline number of nephrologist's office visits at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline number of nephrologist's office visits and the ones at 6 and 12 months will be performed. Data will be extracted from the data flows of healthcare information systems
Change from baseline Dialyzer clearance of urea multiplied by dialysis time and normalized for urea distribution volume (Kt/V) at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline Kt/V and the one at 6 and 12 months will be performed. Data will be extracted from the Tests Laboratory data flows
Change from baseline Estimated Glomerular Filtration Rate (eGFR) at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline eGFR and the one at 6 and 12 months will be performed. Data will be extracted from the Tests Laboratory data flows
Change from baseline Hb at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline Hb and the one at 6 and 12 months will be performed. Data will be extracted from the Tests Laboratory data flows
Change from baseline Ca/P at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline Ca/P and the one at 6 and 12 months will be performed. Data will be extracted from the Tests Laboratory data flows
Change from baseline Parathyroid hormone (PTH) levels at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline PTH and the one at 6 and 12 months will be performed. Data will be extracted from the Tests Laboratory data flows
Change from baseline Average weight loss in HD/PD at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline Average weight loss in HD/PD and the one at 6 and 12 months will be performed. Data will be extracted from the patients' clinical health record
Change from baseline Weight at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline Weight and the one at 6 and 12 months will be performed. Data will be extracted from the patients' clinical health record
Change from baseline HD complications at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline Intratreatment and Extra treatment HD complications and the ones at 6 and 12 months will be performed. Data will be extracted from the patients' clinical health record
Change from baseline PD complications at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline Intratreatment and Extra treatment HD complications and the ones at 6 and 12 months will be performed. Data will be extracted from the patients' clinical health record
Change from baseline Total number of prescribed drugs at 6 and 12 months | Baseline, 6 months and 12 months
  A comparison among the baseline Total number of prescribed drugs and the one at 6 and 12 months will be performed. Data will be extracted from the patients' clinical health record
Change from 6 months Satisfaction score of the system at 12 months (5-level scale) | 6 months and 12 months
  A comparison between the overall satisfaction rating of the system at 6 and 12 months will be carried out.
  A 5-level scale is used (interval scale: 1 to 5): 1=Very Unsatisfied, 2= Unsatisfied, 3=Neutral, 4=Satisfied, 5=Very Satisfied.
  Information collected through a specific questionnaire.
Change from 6 months Usability index of the system at 12 months | 6 months and 12 months
  A comparison between the Usability rating of the whole system and of the individual devices at 6 and 12 months will be carried out. Information collected through a specific questionnaire.
Change from 6 months Time acceptability index at 12 months | 6 months and 12 months
  A comparison between the Patients' acceptance of the time required for the system daily usage at 6 and 12 months will be carried out. Information collected through a specific questionnaire.
Change from 6 months Acceptance of a potential systematic usage at 12 months | 6 months and 12 months
  A comparison between the Patients' acceptance of a potential systematic usage of the system at 6 and 12 months will be carried out. Information collected through a specific questionnaire.
Total number of measurements (systolic blood pressure, pulse rate, oxygen saturation, temperature, weight, electrocardiogram, bio-electrical impedance analysis) | 12 months
  Total number of measurements (systolic blood pressure, pulse rate, oxygen saturation, temperature, weight, electrocardiogram, bio-electrical impedance analysis) performed by patients through the devices he is equipped with.
  Data will extracted from the system service platform.
Total number of measurements (systolic blood pressure, pulse rate, oxygen saturation, temperature, weight, electrocardiogram, bio-electrical impedance analysis) per patient | 12 months
  Total number of measurements performed by each patient through the devices he is equipped with.
  The measurements include the following parameters: systolic blood pressure, pulse rate, oxygen saturation, temperature, weight, electrocardiogram, bio-electrical impedance analysis parameters.
  Data will extracted from the system service platform.
Total number of measurements per parameter (systolic blood pressure, pulse rate, oxygen saturation, temperature, weight, electrocardiogram, bio-electrical impedance analysis) | 12 months
  Total number of measurements per parameter (systolic blood pressure, pulse rate, oxygen saturation, temperature, weight, electrocardiogram, bio-electrical impedance analysis) performed by patients through the devices he is equipped with.
  Data will extracted from the system service platform.
Total number of measurements per parameter (systolic blood pressure, pulse rate, oxygen saturation, temperature, weight, electrocardiogram, bio-electrical impedance analysis) per patient | 12 months
  Total number of measurements per parameter (systolic blood pressure, pulse rate, oxygen saturation, temperature, weight, electrocardiogram, bio-electrical impedance analysis) performed by each patient through the devices he is equipped with.
  Data will extracted from the system service platform.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Bianchi, MD, Study Chair — Azienda Sanitaria Nord Ovest Toscana Italy
Locations (1):
- Azienda Sanitaria NordOvest Toscana, Livorno, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young A, Orchanian-Cheff A, Chan CT, Wald R, Ong SW. Video-Based Telemedicine for Kidney Disease Care: A Scoping Review. Clin J Am Soc Nephrol. 2021 Dec;16(12):1813-1823. doi: 10.2215/CJN.06660521. Epub 2021 Dec 7. PMID 36630403
- [Background] Lindeboom L, Lee S, Wieringa F, Groenendaal W, Basile C, van der Sande F, Kooman J. On the potential of wearable bioimpedance for longitudinal fluid monitoring in end-stage kidney disease. Nephrol Dial Transplant. 2022 Oct 19;37(11):2048-2054. doi: 10.1093/ndt/gfab025. PMID 33544863
- [Background] Gc VS, Iglesias CP, Erdem S, Hassan L, Peek N, Manca A. Using discrete-choice experiments to elicit preferences for digital wearable health technology for self-management of chronic kidney disease. Int J Technol Assess Health Care. 2022 Oct 26;38(1):e77. doi: 10.1017/S0266462322003233. PMID 36286261